CLINICAL TRIAL: NCT07390266
Title: A Randomized, Triple-blind, Placebo-controlled, Cross-over Clinical Trial to Determine the Safety and Efficacy of an Origin Satiety Complex on Self-reported Hunger and Satiety in Healthy Adults
Brief Title: A Clinical Trial to Determine the Safety and Efficacy of an Origin Satiety Complex on Self-reported Hunger and Satiety in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vora Life LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25VRLCR01
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: High BMI; Hunger; Satiety; Healthy Adults
Keywords: Vora Life; Origin Satiety Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Origin Satiety Complex (Experimental): Origin Satiety Complex consists of a mix of L-glutamine, fiber blend, spinach whole herb extract, sweet potato powder, blueberry fruit extract, green coffee bean extract, cinnamon bark extract, and a probiotic blend.
  Interventions: Dietary Supplement: Origin Satiety Complex
- Placebo (Placebo Comparator): Placebo consists of a commercially available juice powder, Tang.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Origin Satiety Complex — Participants will be instructed to consume five doses of study product premixed in 10 ounces of water in an opaque container.
  Arms: Origin Satiety Complex
Other: Placebo — Participants will be instructed to consume five doses of study product premixed in 10 ounces of water in an opaque container.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to the safety and efficacy of the investigational product (IP), Origin Satiety Complex, on hunger and satiety in healthy adults. The main question it aims to answer is what is the difference in the net incremental area under the curve (niAUC) for self-reported postprandial hunger and satiety (T = 0 - T = 10.5 h), as assessed by satiety and hunger items of the Eating Behavior Visual Analog Scales (VAS), between the IP and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males & females 21 - 50 years of age, inclusive
2. BMI between 18.5 - 29.9 kg/m²
3. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
4. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
5. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
6. Agrees to consume the standardized dinner the night prior to study visits and comply with fasting requirements
7. Agrees to avoid alcohol consumption in the 24 hours prior to clinic visits and caffeine consumption and physical exercise on the morning of each study visit
8. Provided voluntary, written, informed consent to participate in the study
9. Healthy as determined by medical history as assessed by the Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of investigational product, placebo, or standardized meal ingredients
3. Poor venous access as assessed by the QI
4. Following a specific diet (e.g., vegetarian, paleo, ketogenic, carnivore, etc.), as assessed by the QI
5. Unstable metabolic disease or chronic diseases as assessed by the QI
6. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
7. Current or history of eating disorders or restricted eating as assessed by the QI
8. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3)
9. Type I or Type II diabetes
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Gastric bypass surgery or other surgeries to induce weight loss
15. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
16. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
17. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
18. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
19. Self-reported confirmation of hypercalcemia and/or hypercalciuria diagnosis, as assessed by the QI
20. Use of medical cannabinoid products
21. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
22. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
23. Alcohol intake average of >2 standard drinks per day as assessed by the QI
24. Alcohol or drug abuse within the last 12 months
25. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the safety and/or efficacy of the investigational product (Sections 7.3.1 and 7.3.2)
26. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
27. Individuals who are unable to give informed consent
28. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The difference in the net incremental area under the curve (niAUC) for self-reported postprandial hunger and satiety | Time (T) 0 to 10.5 hours
  The difference in the net incremental area under the curve (niAUC) for self-reported postprandial hunger and satiety (T = 0 - T = 10.5 h), as assessed by satiety and hunger items of the Eating Behavior Visual Analog Scales (VAS), between the IP and placebo. The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".

SECONDARY OUTCOMES:
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 0 to 1.5 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in fasted state, after a single dose of study product (T = 0 h - T = 1.5 h). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 0 to 5.5 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in a postprandial state, after three doses of study product and two meals (T = 0 h - T = 5.5 ). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 3.5 to 5.5 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in a postprandial state, after three doses of study product and two meals (T = 3.5 h - T = 5.5 h). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 8.5 to 10.5 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in a postprandial state, after five doses of study product and three meals (T = 8.5 h - T = 10.5 h). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 1.5 to 3.75 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in a postprandial state after breakfast and two doses of study product (T = 1.5 h - T = 3.75 h). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 4.5 to 8.5 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in a postprandial state after lunch and four doses of study product (T = 4.5 h - T = 8.5 h). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) between IP and placebo. | 9.5 to 10.5 hours
  The difference in niAUC for self-reported eating behaviors (hunger, fullness, nausea, thirst, amount of food they could eat) as assessed by the Eating Behavior VAS between IP and placebo in a postprandial state after dinner and five doses of study product (T = 9.5 h - T = 10.5 h). The VAS is on a scale of 1 to 10, with 1 being "not hungry at all" and 10 being "extremely hungry".
The difference in self-reported eating behavior (hunger, fullness, nausea, thirst, amount of food they could eat) 90 minutes after each meal | 1.75, 3.75, and 8.75 hours after T0 h
  The difference in self-reported eating behavior (hunger, fullness, nausea, thirst, amount of food they could eat) 90 minutes after each meal as assessed by the Eating Behavior VAS between IP and placebo.
The difference in postprandial glucose between IP and placebo | Baseline and 3, 5, 5.5, and 10 hours
  The difference in postprandial glucose at T = 3, 5, 5.5, and 10 h between IP and placebo
The difference in postprandial glucose between IP and placebo | Baseline and 3, 5, 5.5, and 10 hours
  The difference in postprandial insulin at T = 3, 5, 5.5, and 10 h between IP and placebo
The difference in niAUC(0-10h) for serum glucose between IP and placebo | 0 to 10 hours
  The difference in niAUC(0-10h) for serum glucose between IP and placebo
The difference in niAUC(0-10h) for serum insulin between IP and placebo | 0 to 10 hours
  The difference in niAUC(0-10h) for serum insulin between IP and placebo

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | 0 to 10.5 hours
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in blood pressure (BP) after supplementation | 0 to 10.5 hours
  Clinically relevant changes in blood pressure (BP) after supplementation
Clinically relevant changes in heart rate after supplementation | 0 to 10.5 hours
  Clinically relevant changes in heart rate after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada